CLINICAL TRIAL: NCT02743312
Title: Long-Term Effects of Balance-Based Torso-Weighting: Pilot Study
Brief Title: Long-Term Effects of Torso-Weighting
Acronym: TWPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco State University (Other)
Collaborators: Samuel Merritt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X15-48a
Record Dates: First submitted 2015-10-07; First posted 2016-04-19 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: Balance-Based Torso-Weighting; Physical Activity; Neurorehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Torso Weights then Sham Weights (Experimental): No weights worn for 4 weeks. Garment with torso weights worn 2-4 hours daily for 2 weeks. Then participants cross-over to wear garment with sham weights for 2-4 hours daily for 2 weeks.
  Participants wear the Fitbit Flex throughout.
  Interventions: Device: Torso Weights; Device: Sham Weights; Device: Fitbit Flex
- Sham Weights then Torso Weights (Experimental): No weights worn for 4 weeks. Garment with sham weights worn 2-4 hours daily for 2 weeks. Then participants cross-over to wear garment with torso weights for 2-4 hours daily for 2 weeks.
  Participants wear the Fitbit Flex throughout.
  Interventions: Device: Torso Weights; Device: Sham Weights; Device: Fitbit Flex

INTERVENTIONS:
Device: Torso Weights — Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss.
  Other Names: WT
Device: Sham Weights — Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with sham weights.
  Other Names: SW
Device: Fitbit Flex — Potential effect on participants' physical activity to see their own step count using this wrist-worn remote monitoring device.
  Other Names: remote activity monitoring device

SUMMARY:
The goal of this pilot study is to test the protocol for investigating the longer-term effects of torso weighting on physical activity, number of falls, and muscle activation (when muscles turn on and off and how intensely) in five volunteers with multiple sclerosis. The hypotheses of this study include: torso weighting will (1) increase physical activity, (2) decrease the number of falls, and (3) improve the timing and coordination of muscle activation during balance perturbations.

DETAILED DESCRIPTION:
Torso weighting, using the balance-based torso-weighting (BBTW) method, is an intervention that addresses balance by first challenging stability in standing using a series of perturbations (nudges) and resisted rotations to people. Challenging stability allows the assessor to determine directional instability. Once the direction of instability is determined, small weights are placed on a vest-like garment and retesting of balance occurs. In this study, participants will be tested with no weights (NW), with sham weights (SW), and with BBTW weighting (WT). Following non-weighted baseline assessment, participants will be randomly allocated into the sham weight condition or BBTW weight condition in a cross-over design. The initial condition (NW) will last four weeks and the final two conditions (SW,WT) will last two weeks each. Following each condition, outcome measures will be reassessed. Throughout the study, participants will be asked to wear a commercially-available remote monitoring device (e.g., Fitbit Flex) and keep a daily log of physical activity and number of falls. During the SW and WT conditions, participants will wear the assigned garment for 2-4 hours daily.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported a diagnosis of multiple sclerosis
* Self-reported mild or moderate gait or balance difficulties
* Living in the community rather than in a care facility
* Able to walk independently for at least one minute at a time with or without an assistive device
* No exacerbations within the past 2 months
* Able to get to the testing area and tolerate 2-3 hours of testing for each assessment occasion
* Willing to be nudged by a researcher when standing

Exclusion Criteria:

* Unable to comprehend and follow instructions in English
* Current diagnosis of other neurological disorders such as head injury, stroke, Parkinson disease, or other conditions that affect gait or balance (self-reported)
* Experiencing pain that could be exacerbated by external perturbation while standing
* History of skin reaction to adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Allen, PhD, Principal Investigator — San Francisco State University
Locations (1):
- Samuel Merritt University, Motion Analysis Research Center, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 volunteers were screened for eligibility from November 1, 2015, to April 1, 2016.
Pre-assignment Details: All 5 volunteers were enrolled.
Groups:
- Torso Weights Then Sham Weights: No weights worn for 4 weeks. Garment with torso weights worn 2-4 hours daily for 2 weeks. Then participants cross over to wear garment with sham weights 2-4 hours daily for 2 weeks.
  Participants wear the Fitbit Flex throughout.
  Balance-Based Torso-Weighting (WT): Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with actual weights (but assessors and patients are not told which weights are placed).
  Fitbit Flex: Potential effect on participants' physical activity to see their own step count using this wrist-worn remote monitoring device.
- Sham Weights Then Torso Weights: No weights are worn for 4 weeks. Garment with sham weights worn 2-4 hours daily for 2 weeks. Then participants cross-over to wear garment with torso weights 2-4 hours daily for 2 weeks.
  Participants wear the Fitbit Flex throughout.
  Sham Weights (SW): Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with sham weights (assessors and patients are not told which weights are placed).
  Fitbit Flex: Potential effect on participants' physical activity to see their own step count using this wrist-worn remote monitoring device.
Period: Overall Study
Arm/Group | Torso Weights Then Sham Weights | Sham Weights Then Torso Weights
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Torso Weights Then Sham Weights: No weights worn for 4 weeks. Garment with torso weights worn 2-4 hours daily for 2 weeks. Then participants cross-over to wear garment with sham weights for 2-4 hours daily for 2 weeks.
  Participants wear the Fitbit Flex throughout.
  Torso Weights: Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with actual weights (but the assessors and patients do not know which weights are placed).
  Sham Weights: Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with sham weights.
  Fitbit Flex: Potential effect on participants' physical activity to see their own step count using this wrist-worn remote monitoring device.
- Sham Weights Then Torso Weights: No weights worn for 4 weeks. Garment with sham weights worn 2-4 hours daily for 2 weeks. Then participants cross-over to wear garment with torso weights for 2-4 hours daily for 2 weeks.
  Participants wear the Fitbit Flex throughout.
  Sham Weights: Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with sham weights (but the assessors and patient do not know which weights are placed).
  Torso Weights: Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with actual weights.
  Fitbit Flex: Potential effect on participants' physical activity to see their own step count using this wrist-worn remote monitoring device.
- Total: Total of all reporting groups
Arm/Group | Torso Weights Then Sham Weights | Sham Weights Then Torso Weights | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Steps Per Day
Description: Continuous activity data collection via commercially-available remote monitoring device and stored on server.
Time Frame: up to 8 weeks
Population: Server where data were stored failed. No data analyzed for any participant.
Groups:
- Torso Weights: Garment with torso weights worn 2-4 hours daily for 2 weeks.
  Torso Weights: Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss.
- Sham Weights: Garment with sham weights worn 2-4 hours daily for 2 weeks.
  Sham Weights: Following assessment of an individual's directional instability, small weights are applied to a vest-like garment to correct balance loss. The garment is then taken by another investigator and the actual weights are replaced with sham weights.
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Sensory Organization Test
Description: balance tested during 6 conditions on Neuro-com forceplate and surround and reported as a composite score (across the six conditions), 0-100, with higher scores indicating better balance; measure reported reflects change in the composite score from the visit that initiates Torso-weighting (TW) or sham weights (SW) to the visit that concludes daily wearing of TW or SW
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Torso Weights: Average change in variable from beginning to end of 2 weeks of torso weights.
- Sham Weights: Average change in variable from beginning to end of 2 weeks of sham weights.
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
scores on a scale | 7.4 (8.4) | 1 (9.7)

3. Secondary Outcome: Gait Velocity
Description: As measured using instrumented gait mat.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
meters/second | .125 (.14) | -.03 (.14)

4. Secondary Outcome: Movement Ability Measure, Computer Adaptive Test Version (MAM-CAT)
Description: Online self-report of perceived current movement ability and preferred movement ability. The scores are reported in standardized logits, 0-6, where 6 is competitive level athletic movement. The reported values are the average change in current movement ability from initiation of daily wear to after 2 weeks of daily wear of TW or SW.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
units on a scale | .36 (1.8) | .3 (.7)

5. Secondary Outcome: Activities-Specific Balance Confidence Scale
Description: Self-report measure of perception of confidence under various balance challenges on a scale of 0-100 with 100 being fully confident that the individual can perform the listed balance challenge without falling. Data reported reflect the difference in scores from initiation to the 2-week point after initiation of TW or SW.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Torso Weights: Garment with torso weights worn 2-4 hours daily for 2 weeks.
- Sham Weights: Garment with sham weights worn 2-4 hours daily for 2 weeks.
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
units on a scale | 1.5 (6.6) | 3 (6.9)

6. Secondary Outcome: Multiple Sclerosis Impact Scale 29
Description: Self-report measure of the impact of MS on activities and participation. The scale is reported in a physical and psychological subscale, with higher numbers (out of 100) indicating worse impact of multiple sclerosis (MS) on function. Data are reported as change from initiation of TW or SW to end of 2 weeks of daily wear.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
units on a scale
  Physical score | -6.7 (4.7) | -5.25 (10.5)
  Psychological score | -4.4 (12.2) | -6.1 (10.3)

7. Secondary Outcome: Multiple Sclerosis Walking Scale 12
Description: Self-report measure of the effect of MS on walking ability. Larger numbers out of 100 mean that MS limits walking much more. Data are reported as change in score from initiation of TW or SW to the visit after 2 weeks of daily wear of TW or SW.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
units on a scale | -7.9 (9.6) | -0.8 (13.3)

8. Secondary Outcome: Six-Minute Walk Test
Description: distance participant walks in 6 minutes. Larger numbers indicate more distance covered. Data reported are the change in distance walked from initiation of TW or SW to after 2 weeks of daily wear.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: meters walked
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
meters walked | 47.4 (52) | -19 (44.3)

9. Secondary Outcome: Stride Length
Description: As measured using instrumented gait mat.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
meters | .09 (.09) | -.02 (.11)

10. Secondary Outcome: Percent of Gait Cycle in Single Limb Support
Description: As measured in percent (e.g., 0.35) of gait cycle spent on one limb using instrumented gait mat.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: percentage of gait cycle on one limb
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
percentage of gait cycle on one limb | .0067 (.0062) | -.0026 (.0072)

11. Secondary Outcome: Step Width
Description: As measured using instrumented gait mat.
Time Frame: change from initiation to 2-weeks after initiation of daily wearing of TW or SW
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
meters | -.0084 (.03) | .014 (.014)

12. Secondary Outcome: Electromyography to Assess Muscle Activation
Description: Recording of muscle activation during quiet and perturbed standing before and after intervention at weeks 4, 6, and 8. Average values with and without weighting during each visit.
Time Frame: Week 4, Week 6, Week 8
Population: timing and marker difficulties along with equipment malfunction at some visits resulted in data that could not be analyzed.
Groups:
- No Weights: Vest-like garment is worn for testing during each visit (at 4 weeks, 6 weeks, and 8 weeks) before torso-weights are applied.
Arm/Group | Torso Weights | No Weights
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Falls Recorded in 2 Weeks of Wear Time.
Description: Daily log manually recorded by participant for the 2 weeks of wear time. This is a descriptive measure recording the total count (number) of falls per arm.
Time Frame: count of number of falls recorded at the end of two weeks of wearing TW or SW
Population: total falls in each arm
Measure: Number; unit: falls
Groups:
- Torso Weights: From beginning to end of 2 weeks of daily wearing of torso weights.
- Sham Weights: From beginning to end of 2 weeks of daily wearing of sham weights.
Arm/Group | Torso Weights | Sham Weights
Number analyzed (Participants) | 5 | 5
falls | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months, beginning to end of data collection of any participant
Groups:
- Pre-weighting (no Weights): 4 week baseline period in which participants wore activity monitor but had no other intervention.
Arm/Group | Torso Weights | Sham Weights | Pre-weighting (no Weights)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No